CLINICAL TRIAL: NCT04118322
Title: The Effect of Peppermint Oil on Nausea, Vomiting and Retching in Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Trial
Brief Title: The Effect of Peppermint Oil on Nausea, Vomiting and Retching in Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nuriye EFE ERTÜRK, PhD. Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/72
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Chemotherapy Effect; Adverse Effect; Nursing Caries
Keywords: Aromatherapy; Chemotherapy; Nausea-Vomiting; Nursing; Peppermint Oil
MeSH Terms: interventions — Aromatherapy; peppermint oil

STUDY DESIGN:
Intervention Model Description: Randomised controlled trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The patients in the intervention group applied peppermint oil (3%) on lips three times a day, during the five days following chemotherapy administration, in addition to the standard antiemetic treatments. The data were collected using a Patient Information Form, Rhodes Index of Nausea, Vomiting and Retching (INVR), Visual Analog Scale (VAS) Patient Nausea Severity Follow-up Form, Patient Watch Chart, and Oil Application Protocol. Besides, patients in the intervention group were questioned thoughts associated with peppermint oil application using individual in-depth interview method.
  Interventions: Other: aromatherapy (peppermint oil)
- control group (No Intervention): The control group underwent only the routine treatment.

INTERVENTIONS:
Other: aromatherapy (peppermint oil) — The patients in the intervention group received routine medical treatment program and were asked to put one drop of peppermint oil upon lips following chemotherapy administration. Before peppermint oil application; the researcher theoretically and practically provided a training of 8-10 minutes about the use of peppermint oil and the patients were requested to apply this oil three times a day according to "Oil Practice Guide" (See Fig. 2) in the morning (09:00), at noon (15:00) and in the evening (21:00).
  Aromatherapy essential oil used was a mixture of English peppermint (Mentha piperita; 3%) and sweet almond oil (30 ml)
  Arms: intervention group

SUMMARY:
The aim of this study was to determine the effect of peppermint oil upon incidence of nausea, vomiting and retching, nause severity, and the usage amount of antiemetics in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Nausea, vomiting and retching symptoms are among the most common adverse effects of chemotherapy and are defined with expressions like "the biggest problem including pain" by patients. Chemotherapy-induced nausea and vomiting (CINV)' is reported leads to fluid-electrolyte imbalance, dehydration, loss of weight, physiological effects caused by poor drug absorption or decreased elimination from kidneys as well as negative effects in one's social life, work-life, activities of daily life and psychological status. Also, nausea-vomiting may cause some patients to refuse chemotherapy or to discontinue the treatment. Inadequate control of CINV leads patients to integrative health practices.

The study was realized as a randomized controlled study in order to explore the effect of use of 3% peppermint oil applied on lips three times a day during the five days following chemotherapy upon incidence nausea, vomiting, and retching, nausea severity and quantity use of antiemetics in cancer patients undergoing chemotherapy.The study was initiated on the 10.09.2017 and in this study were interviewed with 250 patients. 90 patients that met inclusion criteria were contacted. The study was completed with 36 intervention patients and with 44 control patients (See Fig. 1). For determine to sample size, while patients were being allocated to the study groups, post hoc power analysis was periodically done with the data obtained. The sample size for this study was calculated using the MedCalc (32-bit). The process continued until the necessary sample size was reached. According to power analysis, α = 0.05 and β =0.20, and the power of the study was 99.9%.

Randomization In order to provide randomization was preferred ballot method. As a result of the ballot, the first patient who inclusion criteria of study was allocated to the intervention group while the next one to the control group. After participant enrollment, patients were assigned to the two groups in a 1:1 ratio according to this rule. Because of it is not known whether nausea/vomiting experience of patients who first time chemotherapy receiving, study groups included patients receiving two or more chemotherapy.

Interventions 2.4.1. The control group The control group underwent only the routine treatment. The patients in the control group, Patient Watch Chart, Patient Nausea Severity Follow-up Form, and INVR, marked by patients and They were returned the duly completed these forms to the researcher when they came to hospital for the next chemotherapy treatment. Patient Watch Chart, and INVR skala of patients who illiterate were filled in by the pollster, according to expression of patient. In order to fill in Patient Watch Chart, and INVR phone interviews were made twice a day (morning-evening) by the pollster and the participants at a suitable time determined together.

2.4.2. Intervention group The patients in the intervention group received routine medical treatment program and were asked to put one drop of peppermint oil upon lips following chemotherapy administration. Before peppermint oil application; the researcher theoretically and practically provided a training of 8-10 minutes about the use of peppermint oil and the patients were requested to apply this oil three times a day according to "Oil Practice Guide" (See Fig. 2) in the morning (09:00), at noon (15:00) and in the evening (21:00). The mobile phones of the participants were set to these hours and the alarm system continued in this manner for five days. The participants whose mobile phones were not set to these hours were called by the researcher in order to recall them of the protocol. Before peppermint oil application, Patient Opinion Form (pre-application) were asked to the participants and their answers were written down. Similarly; after peppermint oil application, same form (post-application) were asked and the answers were written down. Patient Watch Chart, Patient Nausea Severity Follow-up Form, and INVR, marked by patients and They were returned the duly completed these forms to the researcher when they came to hospital for the next chemotherapy treatment. Patient Watch Chart, and INVR skala of patients who illiterate were filled in by the pollster, according to expression of patient. In order to fill in Patient Watch Chart, and INVR phone interviews were made twice a day (morning-evening) by the pollster and the participants at a suitable time determined together.

Patients in the intervention and control groups were allowed to take standard antiemetic medications and other drugs taken for different medical problems during and after the day of peppermint oil application. As a part of standard antiemetic treatment; patients were given " in isotonic solution 5-HT3 receptor antagonists (palonosetron, granisetron (Kytril))+ steroids (dexamethazon (Decort)) + antihistaminic (Avil or Systral ampul) + Metpamid ampul" before chemotherapy.

Onzyd 8 mg (ondansetron) + metpamid tb. has been prescribed by oncologist, for able to use at patient's home.

ELIGIBILITY:
Inclusion Criteria: Patients who

* were aged ≥18 years,
* were able to understand Turkish language and to communicate in Turkish language,
* had cancer diagnosis,
* received chemotherapy treatment for -at least- the second time with similar chemotherapeutic agents,
* experienced nausea symptoms according to VAS
* were not pregnant and not intending pregnancy,
* had -at most- stage III cancer
* presented no psychiatric disorders,
* were not included in pre-implementation phase of the study were accepted to the study.

Exclusion Criteria:Patients who

* suffered from another disease that may affect nausea vomiting status,
* were allergic to or disturbed by smell of peppermint,
* were newly diagnosed, and receiving chemotherapy for the first time,
* received concomitant radiotherapy,
* received other complementary and integrative health practices during the treatment were not accepted to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 1 day (first day)
  The form was consisted of 17 statements in order to explore patients' socio-demographic characteristics (age, sex, educational status, marital status, number of children, etc.), and diagnosis, treatment protocol, and complementary and integrative health practices used to cope with cancer and nausea-vomiting symptoms.
Visual Analog Scale (VAS)- Nausea Severity | 1 day (fist day)
  The scale (VAS) was used to accept patients to the study. VAS is composed of 10-cm (100 mm) line which at the left end by words "No nausea 0" and increased numbers indicated rising nause levels; at the right end "Severe nausea 10". The patient is asked to place a mark on the scale to indicate the level of intensity of his or her nausea. Distance of patient's mark to left end is measured with a ruler in millimeter and is accepted and written as score

SECONDARY OUTCOMES:
Patient Watch Chart | 1-5 days
  The form was separately designed for the intervention and control groups after a thorough review of the relevant literature. Patient Watch Chart was designed to explore status of use of antiemetics prescribed only by physicians for the patients in the control group while in the intervention group, to explore status of use of antiemetics and status of peppermint oil.
The Index of Nausea, Vomiting, and Retching- INVR | 1-5 days
  The index was developed by Rhodes V. and Mc Daniel R. (Rhodes & Mc Daniel, 1999) in order to explore post chemotherapy nausea, vomiting, and retching frecuency and distresses that patients experience. The index is composed of 8 questions. Assign a numeric value to each response from 0, (the least amount of distress), to 4, (the most distress). Total symptom experience from nausea and vomiting is calculated by summing the patient's responses to each of the eight items on the Rhodes INV. The potential range of scores is from a low of 0 to a maximum of 32. Patients are required to fill in the form in the most suitable period of 12 hours that they decide. There are three subdimensions: symptoms experience, symptoms occurrence, and symptoms distress. In order to score the INVR; 1st, 3rd, 6th and 7th items should be reversed.
Peppermint Oil Application Protocol | 1-5 days
  The guideline were prepared in line with expert opinion and literature in order to show stages and important oints of oil application and to make sure that the oil application would be carried out in the same manner by all the patients. The aromatherapy essential oil used was a mixture of English peppermint (Mentha piperita; 3%) and sweet almond oil (30 ml), Patients were informed of keeping the aromatic mixture in a closed and dark bottle, in a cool place and away from sunshine. The peppermint oil application was carried out according to Oil Practice Guide (See Fig. 2) by the patients in the intervention group.
Patient Opinions Form of Peppermint Oil Application | only 1st and 5th day
  The form included semi-structured questions designed in line with expert opinions and literature in order to identify opinions of the patients in the intervention group about the peppermint oil application (Muz & Taşcı, 2017). The questions in the form were asked to the patients before and after peppermint oil application and patient opinions were voice-recorded or written down. Before peppermint oil application; the questions ("What do nausea and/or vomiting mean for you?, How do these symptoms influence your life?, Do you believe that the oil to be used will help lessen your symptoms?") were asked whereas after peppermint oil application; the questions ("Do you think that peppermint oil application has had effect upon nausea, vomiting, and retching symptoms?, How has peppermint oil application affected your daily life?, What are the easy and difficult sides of peppermint oil application?") were asked to explore patient views.
VAS-Patient Nausea Severity Follow-up Form | 1-5 days
  In order to assess severity of nausea experienced by patients after chemotherapy administration; VAS- Patient Nausea Severity Follow-up Form was developed by the researcher and marked by the patients in intervention group and control group. The form consists of VASs that marked two times a day -in the morning and in the evening- during five days (Zorba & Özdemir, 2018; Arslan & Özdemir, 2015). Marking and evaluation of the VAS's in the form were done according to the principles in the Visual Analogue Scale (VAS) - Severity of Nausea.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuriye EFE ERTURK, Batman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lua PL, Salihah, Mazlan N. Effects of inhaled ginger aromatherapy on chemotherapy-induced nausea and vomiting and health-related quality of life in women with breast cancer. Complementary Therapies in Medicine 23: 396-404, 2015 https://doi.org/10.1016/j.ctim.2015.03.009. Zorba,P,Özdemir L. The preliminary effects of massage and inhalation aromatherapy on chemotherapy-induced acute nausea and vomiting. Cancer Nursing 41(5): 359-366, 2018 https://doi.org/10.1097/NCC.0000000000000496. Seale MK. The Use of Peppermint Oil to Reduce the Nausea of the Palliative Care and Hospice Patient [dissertation]. Boiling Springs, NC: School of Nursing, Gardner-Webb University.2012 Arslan M, Özdemir L. Oral intake of ginger for chemotherapy-induced nausea and vomiting among women with breast cancer. Clinical Journal of Oncology Nursing 19(5): E92-97, 2015 http://doi.org/10.1188/15.CJON.E92-E97. Muz G Taşcı S. Effect of aromatherapy via inhalation on the sleep quality and fatigue level in people undergoing hemodialysis. Applied Nursing Research, 37, 28-35, 2017 http://dx.doi.org/10.1016/j.apnr.2017.07.004. Rhodes V, Mc Daniel R. The index of nausea, vomiting and retching: A new format of the index of nausea and vomiting. Oncology Nursing Forum 26(5): 889-894, 1999.